CLINICAL TRIAL: NCT07135375
Title: Postoperative Rotator Cuff: Functional, Pain and Sleep Quality
Brief Title: Postoperative Rotator Cuff Rehabilitation: Functional, Pain and Sleep Quality
Acronym: REHAB-PSF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LAURA CASTILLO VEJAR (Other)
Responsible Party: Sponsor-Investigator, LAURA CASTILLO VEJAR, Sponsor- Principal investigador, Physiotherapist, TRIMEDKINE
Organization: TRIMEDKINE (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N°1
Record Dates: First submitted 2025-07-30; First posted 2025-08-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Injuries; Functionality; Pain; Sleep; Rehabilitation; Rotator Cuff
Keywords: Rehabilitation; Rotator cuff
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study using non probability convenience sampling
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard protocol (Active Comparator): According American Society of Shoulder and elbow therapist
  Interventions: Other: Rehabilitation protocol
- Modified protocol (Experimental): According to the number of tendons treated
  Interventions: Other: Rehabilitation protocol

INTERVENTIONS:
Other: Rehabilitation protocol — The modified protocol will be implementen based on available scientific evidence and guided by the consensus remaches with the traumatologist at the physiotherapy center

SUMMARY:
Rotator cuff injuries are the third leasing cause of pain and disability, accounting for 16% of all musculoskeletal injuries. Following surgical intervention, patients typically undergo a 4 to 6 week immobilization period before starting physical therapy. This rehabilitation phase can last between 4 to 6 months. Despite this, there is currently a lack of clear guidelines regarding specific physical therapy protocols or the expected post surgical recovery for patients who have undergone rotator cuff repair.

DETAILED DESCRIPTION:
Objective: To compare the effectiveness of a differentiated rehabilitation protocol based on the number of tendons repaired versus a standard rehabilitation protocol, regarding functionality, pain, subjective perception of sleep quality, and mobility, in patients who have undergone surgical rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* People over 50 years of age
* People have undergone arthroscopic rotator cuff of one or more tendons.
* Patients must sign informed consent and undergo physical therapy center (up to week 12 postoperatively).

Exclusion Criteria:

* Patients who develop postoperative stiffness or adhesive capsulitis during the rehabilitation process.
* Patients with symptoms of cervical radiculopathy or previously diagnosed sleep disorders.
* Patients with neurological or cognitive disorders who have difficulty following instructions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Functionality | 3,6,9 and 12 weeks postoperatively
  QuickDash questionnaire will be administered, which provides information on the level of shoulder disability. The results of this questionnaire are reported as a percentage ranging from 0 to 100%. The higher the score, the greater the level of disability.
Pain nocturnal, dynamic and static | 3,6,9 and 12 weeks postoperatively
  Numeric visual scale, considering 0 as no pian and 10 as the maximum perceived pain. The patient will be asked about his pain at rest, movement, and at night.
Sleep quality | 3,6,9 and 12 weeks postoperatively
  Subjective perception of sleep quality was assessed through questions regarding hours of sleep, number of times awakened due to pain, and use of medication to control nigth time sleep.

SECONDARY OUTCOMES:
Range of movility | 3,6,9 and 12 weeks postoperatively
  The movement of flexion, abduction, internal and external rotation of the shoulder are evaluated by means of goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Laura LA Castillo-Vejar, Principal Investigator — TRIMEDKINE
Locations (2):
- Chile (2):
  - Temuco, senador estebanez 779, Temuco
  - Trimedkine, Temuco

IPD SHARING:
Plan to Share IPD: Yes
Participant information that supports the publicación results
Supporting Information: Study Protocol, SAP
Time Frame: The proceso is complete
Access Criteria: Online